CLINICAL TRIAL: NCT06245460
Title: Evaluation by Ultrasound Imaging of Local Anesthetic Spread to the Popliteal Fossa During an Adductor Canal Block
Acronym: EchoCAdd
Status: Terminated | Type: Observational
Why Stopped: Principal investigator want to stop the study then begining another new one
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP231771; 2023-A01774-41 (Registry Identifier: IDRCB)
Record Dates: First submitted 2024-01-30; First posted 2024-02-07 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Knee Injuries
Keywords: knee surgery; ultrasound; analgesia; pain
MeSH Terms: conditions — Knee Injuries; Agnosia; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Adductor canal block is an effective analgesic technique for major knee surgery. However, the saphenous nerve block is not sufficient to explain this block's efficiency. It has been shown that adductor canal block can spread to the tibial and fibular nerves through the adductor hiatus. However this diffusion's frequency has never been measured. The main objective of this study is to assess the frequency of the spread of the adductor canal block to the fibular and tibial nerves assessed by ultrasound observation at the popliteal fossa.

DETAILED DESCRIPTION:
Adductor canal block is an effective analgesic technique for major knee surgery. The PROSPECT group recommends this block in first intention for locoregional anesthesia in total knee arthroplasty. It has been shown to not be inferior to femoral nerve block in this indication.

The adductor canal block targets the saphenous nerve and, through its spread in the adductor canal, the posterior branch of obturator nerve and the vastus medialis nerve. However these nerves can't fully explain this block's efficiency.

It has been shown that local anesthetic can spread in the adductor canal to the tibial and fibular nerves through the adductor hiatus. However, this spread is inconstant, and no study has evaluated the frequency of this spread yet.

The main objective of this study is to assess the diffusion's frequency of adductor canal block to fibular and tibial nerves through ultrasound observation at the popliteal fossa.

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective knee surgery under general anesthesia
* in center of Ambroise Paré hospital
* receiving an adductor canal block

Exclusion Criteria:

* patients cognitively impaired
* patients suffering from peripheral neuropathy at the lower limb
* patients receiving an IPACK block or surgical knee infiltration to complete the adductor canal block analgesia
* patients who refused to take part in this study
* pregnant or breastfeeding patients
* patients under guardianship
* imprisoned patients
* patients without any medical insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will be all the consecutive patients scheduled for elective knee surgery under general anesthesia in our center and receiving an adductor canal block.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2024-03-05 (Actual); Primary Completion 2025-04-08 (Actual); Study Completion 2025-04-08 (Actual)

PRIMARY OUTCOMES:
Frequency of local anesthetic's spread | at baseline
  The primary outcome is the frequency of local anesthetic's spread to tibial and fibular nerve during an adductor canal block, assessed by ultrasound imaging at the popliteal fossa level. The ultrasound images will be recorded and then assessed by two independent anesthesiologists.

SECONDARY OUTCOMES:
Frequency of altered sensibility | at one and four hours
  Frequency of altered sensibility and motricity in fibular and tibial nerves territories assessed at one and four hours after the adductor canal block has been performed.
Correlation between local anesthetic spread and clinical alteration | at baseline, hour 1 and hour 4th
  Correlation between local anesthetic spread to tibial and fibular nerves during adductor canal block assessed by ultrasound imaging and clinical alteration of sensibility and motricity in these nerves' territories.

CONTACTS AND LOCATIONS:
Overall Officials: Romuald Henry, MD, Principal Investigator — Department of anesthesia, Ambroise Paré Hospital - APHP
Locations (1):
- Department of anesthesia, Ambroise Paré Hospital - APHP, Boulogne-Billancourt, France